CLINICAL TRIAL: NCT01846585
Title: The Effectiveness of Non-Pharmacological Treatment for Insomnia During Pregnancy
Brief Title: Treatment for Insomnia During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rachel Manber, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23501; R01NR013662-01 (NIH)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABTI (Other): Arousal Based Therapy for Insomnia
  Interventions: Behavioral: Arousal Based Therapy for Insomnia
- CBTI (Other): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Arousal Based Therapy for Insomnia — Intervention includes education about sleep and a desensitization technique to reduce sleep interfering arousal
  Arms: ABTI
Behavioral: Cognitive Behavioral Therapy for Insomnia — Intervention includes education about sleep and behavioral and cognitive strategies to improve sleep
  Arms: CBTI

SUMMARY:
The aim of the study is to improve sleep during pregnancy and the postpartum period in women who are experiencing insomnia, using a brief non-pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual (IV-TR edition) criteria for insomnia (duration criterion - 1 month)
* Pregnant with gestational age between 18-32 weeks.
* Adequately fluent in English or Spanish.

Exclusion Criteria:

* Some co-morbid sleep disorders (e.g., moderate to severe obstructive sleep apnea)
* Co-morbid psychiatric disorder
* Use of medications, herbs or other drugs with known effects on sleep
* Unstable medical conditions
* Currently engaged in psychotherapy or other treatments for insomnia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Rate of insomnia remission | Baseline to 30 weeks postpartum

SECONDARY OUTCOMES:
Insomnia severity | Baseline to 30 weeks postpartum
Depression severity | Baseline to 30 weeks postpartum
Sleep Characteristics | Baseline to 30 weeks postpartum
  Self-report measures characterizing sleep onset latency (time to fall asleep), wake after sleep onset, sleep duration.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Manber, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Manber R, Bei B, Suh S, Simpson N, Rangel E, Sit A, Lyell DJ. Randomized controlled trial of cognitive behavioral therapy for perinatal insomnia: postpartum outcomes. J Clin Sleep Med. 2023 Aug 1;19(8):1411-1419. doi: 10.5664/jcsm.10572. PMID 37078188
- [Derived] Badon SE, Dietch JR, Simpson N, Lyell DJ, Manber R. Daytime napping and nighttime sleep in pregnant individuals with insomnia disorder. J Clin Sleep Med. 2023 Feb 1;19(2):371-377. doi: 10.5664/jcsm.10350. PMID 36448328
- [Derived] King LS, Rangel E, Simpson N, Tikotzky L, Manber R. Mothers' postpartum sleep disturbance is associated with the ability to sustain sensitivity toward infants. Sleep Med. 2020 Jan;65:74-83. doi: 10.1016/j.sleep.2019.07.017. Epub 2019 Jul 27. PMID 31734620
- [Derived] Manber R, Bei B, Simpson N, Asarnow L, Rangel E, Sit A, Lyell D. Cognitive Behavioral Therapy for Prenatal Insomnia: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):911-919. doi: 10.1097/AOG.0000000000003216. PMID 30969203